CLINICAL TRIAL: NCT05158010
Title: Advancing Tools for Human Early Lifecourse Exposome Research and Translation- Adolescence Follow-up of the HELIX Subcohort
Acronym: ATHLETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A03533-36
Record Dates: First submitted 2021-03-19; First posted 2021-12-15 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Exposure; Health Behavior; Environment
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HELIX's follow-up (Other)
  Interventions: Other: HELIX's follow-up

INTERVENTIONS:
Other: HELIX's follow-up — * Visit 1 (Day 0): clinical examination (anthropometry, bioimpedance, blood pressure,spirometry), neurodevelopment computer testing, questionnaires (Physical activity,diet, psychological distress, tobacco exposure, pubertal development, sleeping patterns, light exposure before going to sleep, outdoor environment (green spaces, noise), address history, home environment, socio-economic status, noise, psychological distress, medical history, medication use) 7 consecutive days (minimum) of personal exposure monitoring including wearing an actigraph, a Smartphone (GPS data), carrying a NO2 diffusion tube, collection of hair, stool, urines (2 urines during 6 consecutive days) and filling a sleep and physical activity diary
  * Visit 2 (Day 8): blood collection early in the morning and collection of all the 7- days personal monitoring material, and stools and urines samples.

SUMMARY:
ATHLETE will set up a prospective Europe-wide exposome cohort covering the first 2 decades of the life course, which will integrate data on the external, chemical, physical,behavioral, and social domains of the exposome, as well as on health outcomes and biological omics responses, from preconception until adolescence. As part of ATHLETE, the investigators will follow up a unique existing exposome cohort into adolescence (the HELIX Subcohort).

ELIGIBILITY:
Inclusion Criteria:

For the adolescent :

* Subject of the EDEN cohort included in the Helix cohort in 2014-2015 in Poitiers (16-19 years old)
* Subject benefiting from a Social Security scheme or benefiting through a third party

For the person legally responsible :

* The legal guardian, if possible the mother, of the adolescent included in Athlete ;
* Subject benefiting from a Social Security scheme or benefiting through a third person;
* Free subject, without tutorship or guardianship or subordination.

Exclusion Criteria:

* Concomitant participation in another clinical research study.
* Persons not benefiting from a Social Security scheme or not benefiting through a third party.
* Adolescents who are incapable or who do not give their consent to follow the study procedures

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Urinary biomarkers exposure | One week
  Measure of phtalates, phenols, pesticides, (organophosphorus pesticides, metabolites of pyrethroids, 2,4-dichlorophenoxyacid, boscalid, imazalil), cotinine, glycol ethers, polycyclic aromatic hydrocarbon, creatinine, exogenous metabolomics, in a weekly pool of urine collection

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France